CLINICAL TRIAL: NCT00422890
Title: Treatment of Imminent Haematological Relapse in Patients With AML and MDS Following Allogeneic Stem Cell Transplantation With 5-azacitidine (Vidaza®)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: MD Uwe Platzbecker, Dresden University of Technology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TUD-RELAZA-008; 2006-001040-31 (EudraCT Nr.)
Record Dates: First submitted 2007-01-15; First posted 2007-01-17 (Estimated); Last update posted 2011-07-11 (Estimated); Status verified 2011-07

CONDITIONS: Myeloid Leukemia; Myelodysplastic Syndrome
Keywords: Acute myeloid leukaemia or Myelodysplastic syndrome
MeSH Terms: conditions — Leukemia, Myeloid; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute

INTERVENTIONS:
Drug: 5-Azacytidin — in case of decreasing CD34 chimerism

SUMMARY:
Efficacy and safety of 5-Azacytidin in the treatment of the haematological relapse in patients suffering from acute myeloid leukaemia or myelodysplastic syndrome with falling CD34-chimerism after hematopoietic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

Screening phase:

* Age > 18 years
* Patients with CD34+ AML or MDS post-allogeneic HSCT
* Written patient consent after consultation

Treatment phase

* AML/MDS: donor chimerism < 80% in the CD34+ subpopulation following allogeneic HSCT in patients with CD34+ AML or MDS, but with no haematological relapse (blasts < 5% in bone marrow)
* Leukocytes > 3 Gpt/l and platelets > 75 Gpt/l (transfusion-independent)

Exclusion Criteria:

* Known intolerance to 5-azacitidine or mannitol
* Uncontrollable infectious disease
* Patients with active hepatitis B or C or HIV infection
* Severe hepatic function impairment (ASAT and ALAT may not be above three times the normal value) or hepatic cirrhosis, or malignant hepatic tumour
* Renal function impairment (creatinine > twice the normal value, creatinine clearance < 50 ml/min)
* Pregnancy or lactation
* Women of childbearing age, except for those who meet the following criteria:
* postmenopausal (12 months natural amenorrhoea)
* postoperative (6 weeks after bilateral ovarectomy with or without hysterectomy)
* regular and correct use of a contraceptive method with an error rate < 1% per year (e.g. implants, depot injections, combined oral contraceptives, intrauterine device - IUD, whereby hormonal coils with a Pearl Index of < 1% are safer than copper coils)
* sexual abstinence
* Partner vasectomy
* Men who do not use one of the following for contraception:
* sexual abstinence
* post vasectomy
* condoms
* Participation of the patient in a drug trial outside the indication of allogeneic transplantation up to four weeks before study initiation
* Addictive or other illnesses that prevent the person concerned from comprehending the nature and impact, as well as potentical consequences of the clinical trial
* Evidence that the patient may intentionally not comply with the protocol, e.g. lack of cooperation With the exception of a known allergic reaction or intolerance to 5-azacitidine, these criteria do not apply to the screening phase.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2007-01; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Efficacy of 5-Azacytidin in the treatment of the haematological relapse in patients suffering from acute myeloid leukaemia or myelodysplastic syndrome with falling CD34-chimerism after hematopoietic stem cell transplantation. | 4 months

SECONDARY OUTCOMES:
Safety of 5-Azacytidin in the treatment of the haematological relapse in patients suffering from acute myeloid leukaemia or myelodysplastic syndrome with falling CD34-chimerism after hematopoietic stem cell transplantation. | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Platzbecker, MD, Principal Investigator — Univesity Hospital Dresden, department of medicine
Locations (1):
- University hospital Dresden, department of medicine, Dresden, Saxony, Germany

REFERENCES:
- [Derived] Colbers A, Best B, Schalkwijk S, Wang J, Stek A, Hidalgo Tenorio C, Hawkins D, Taylor G, Kreitchmann R, Burchett S, Haberl A, Kabeya K, van Kasteren M, Smith E, Capparelli E, Burger D, Mirochnick M; PANNA Network and the IMPAACT 1026 Study Team. Maraviroc Pharmacokinetics in HIV-1-Infected Pregnant Women. Clin Infect Dis. 2015 Nov 15;61(10):1582-9. doi: 10.1093/cid/civ587. Epub 2015 Jul 22. PMID 26202768